CLINICAL TRIAL: NCT00934414
Title: A Parallel, Controlled, Multi-Center, Single-Dose, One-Period Euglycemic Clamp Study Comparing Prandial Inhalation of Technosphere Insulin in Smokers and Non-Smokers With Type 2 Diabetes
Brief Title: Clamp Study Comparing Inhalation of Technosphere®/Insulin in Smokers and Non-Smokers With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Anders Boss, MannKind Corporation
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MKC-TI-016
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smokers (Experimental)
  Interventions: Drug: Technosphere Insulin Inhalation Powder
- Non-Smokers (Experimental)
  Interventions: Drug: Technosphere Insulin Inhalation Powder

INTERVENTIONS:
Drug: Technosphere Insulin Inhalation Powder — 30U

SUMMARY:
Twelve smoking and twelve non-smoking subjects with Type 2 Diabetes Mellitus will be enrolled in this study to determine the effect of Technosphere® Insulin Inhalation Powder on insulin in the body during a clamp procedure.

DETAILED DESCRIPTION:
MKC-TI-016 is a parallel, prospective, controlled, open-label, 1-period, single-dose trial utilizing a hyperinsulinemic-euglycemic clamp procedure to evaluate the bioavailability and bioeffect of inhaled TI Inhalation Powder in type 2 diabetic subjects who smoke compared to nonsmoking type 2 diabetic subjects.

ELIGIBILITY:
Inclusion Criteria:

* Non Smoking: Clinical diagnosis of type 2 diabetes mellitus.
* Non Smoking: Current basal and prandial insulin therapy for at least 6 weeks either alone or in combination with = 2 OHA
* Non Smoking: Negative urine cotinine test.
* Non Smoking: Non-smoker for at least 2 years.
* Smoking: Clinical diagnosis of type 2 diabetes mellitus.
* Smoking: Have been smoking for at least 5 years
* Non Smoking: Body Mass Index (BMI) of = 40 kg/m2.
* Non Smoking: Glycosylated hemoglobin (HbA1c) of = 12%.
* Non Smoking: If other medications (other than oral anti-diabetic agents) in addition to insulin are taken at screening, the subject must be on a stable regimen as defined by continued use of the same dose of each medication for a period of at least 12 weeks immediately prior to trial enrollment.
* Non Smoking: Forced expiratory volume in one second / forced vital capacity (FEV1/FVC) of = NHANES III predicted Lower Limit of Normal.
* Non Smoking: FVC of = 80% NHANES III predicted value.
* Non Smoking: DLco of = 70% (uncorrected) Miller predicted value.
* Non Smoking: No upper respiratory infections within the last 15 days or lower respiratory infection within the last 30 days.
* Non Smoking: Must be of non-childbearing potential or using adequate birth control measures
* Smoking: Positive cotinine test.
* Smoking: Current basal and prandial insulin therapy for at least 6 weeks either alone or in combination with = oral antihyperglycemic agents.
* Smoking: BMI of = 40 kg/m2.
* Smoking: HbA1c of 12%.
* Smoking: If other medications (other than oral anti-diabetic agents) in addition to insulin are taken at screening, the subject must be on a stable regimen as defined by continued use of the same dose of each medication for a period of at least 12 weeks immediately prior to trial enrollment.
* Smoking: FEV1/FVC = NHANES III Predicted Lower Limit of Normal
* Smoking: FEV1 and FVC of = 60% NHANES III predicted value.
* Smoking: DLco = 70% of (uncorrected) of Miller predicted value.
* Smoking: No upper respiratory infections within the last 15 days or lower respiratory infection within the last 30 days.
* Smoking: Must be of non-childbearing potential or using adequate birth control measures.

Exclusion Criteria:

* Diabetes mellitus type 1.
* Total daily insulin requirement of = 1.4 U/kg.
* Intake of any drug or herbal preparation which, in the evaluation of the Investigator, may interfere with the clinical trial results by causing clinically relevant interference with glucose utilization, insulin action, or recovery from hypoglycemia (eg, systemic corticosteroids, oral or inhaled glucocorticosteroids).
* History of hypersensitivity to the trial drug or to drugs with similar chemical structures.
* Treatment with any investigational drug within 90 days prior to enrollment of trial.
* Progressive fatal disease.
* History of malignancy within five years of trial entry (other than basal cell carcinoma).
* Evidence of severe secondary complications of diabetes (neuropathy, nephropathy as evidenced by creatinine > 1.6 mg/dL for females or > 1.8 mg/dL for males, Stage III or IV retinopathy (according to the MKC diabetic retinopathy scale, see Appendix 1.1 of protocol), or severe peripheral vascular disease).
* Previous history of anaphylaxis or angioedema.
* Evidence of clinically significant autonomic neuropathy (gastroparesis, orthostatic hypotension or hypoglycemia unawareness).
* Myocardial infarction or stroke within the preceding six (6) months.
* Positive hepatitis B (HBsAg) or positive Human Immunodeficiency Virus (HIV) serology or active Hepatitis C (HepCAb) at screening.
* History or presence of clinically significant cardiovascular, hepatic, gastrointestinal, neurological or infectious disorders capable of altering the absorption, metabolism or elimination of drugs, or constituting a significant risk factor when taking trial medication.
* ALT or AST > 3 times the upper limit of the normal reference range.
* Anemia (hemoglobin levels < 11 g/dL for females and < 12 g/dL for males).
* On-going respiratory infection.
* Prior diagnosis of systemic autoimmune or collagen vascular disease requiring previous or current treatment with systemic corticosteroids, cytotoxic drugs, or penicillamine
* Pregnancy, lactation, or the intent of becoming pregnant during the trial period.
* Women of childbearing potential practicing inadequate birth control (adequate birth control is defined as using oral contraceptives, condoms or diaphragms with spermicide, intrauterine devices, or surgical sterilization).
* Current drug or alcohol abuse (regular alcohol intake > 14 units/week), or history which in the opinion of the investigator would not make the subject a suitable candidate for participation in this trial. A unit of alcohol is defined as 8 g of ethanol, ¼ liter of beer or 1 glass of wine or 1 measure of spirits.
* Investigator or site personnel directly affiliated with this trial, and their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-08; Primary Completion 2006-08 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
To compare the relative bioavailability and bioeffect of TI Inhalation Powder in subjects with type 2 diabetes who smoke and who do not smoke to determine relative insulin bioavailability | 15 to 52 days

CONTACTS AND LOCATIONS:
Locations (1):
- Profil Institute for Clinical Research, Chula Vista, California, United States